CLINICAL TRIAL: NCT02514161
Title: Effects of Manual Therapy and Respiratory Muscle Training on the Maximal Inspiratory Pressure in Moderate Smokers
Brief Title: Respiratory Exercises Versus Manual Therapy and Respiratory Exercises in Moderate Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Madrid (Other)
Responsible Party: Principal Investigator, Ibai López-de-Uralde-Villanueva, Principal Investigator, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSEU La Salle
Record Dates: First submitted 2015-07-29; First posted 2015-08-03 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-07

CONDITIONS: Manual Therapies; Respiratory Muscle Training; Exercise Therapy; Inspiratory Capacity
Keywords: Smokers; Maximum Inspiratory Pressure
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inspiratory Muscle Training Group (IMT) (Active Comparator): The IMT program consisted of supervised and domiciliary exercises.
  1. - The supervised exercises was performed in the presence of physiotherapist. This consisted of 30 min 2 days for 4 weeks using the threshold device (Powerbreathe classic level 1, Gaiam Ltd; Southam, Warwickshire, UK). This program involve 5 sets of 5 repetitions with 30 seconds rest between each one. The load of the training was distributed as follow:
     * First week: 30% Maximum Inspiratory Pressure (MIP)
     * Second week: 40% MIP
     * Third week: 50% MIP
     * Fourth week: 60% MIP
  2. - The domiciliary exercises consisted of Yoga Breathing Exercises (Pranayama) that combines the inspiration and expiration through one or both nostrils, and requires the activation of chest and abdomen
  Interventions: Other: Inspiratory Muscle training
- IMT + Manual Therapy and Motor Control Exercises (Experimental): The protocol for this group is identical to the previous group with the sole difference that is added a manual therapy (MT) and a motor control exercises (MCE). The MT protocol was performed for 15min, whereas the MCE was 10min. Below it described both protocols:
  1. - MT:
     * Upper cervical region mobilization in flexion
     * Lower cervical postero-anterior mobilization + maintained traction
     * Costovertebral joint postero-anterior mobilization
     * Thoracic vertebral posteroanterior mobilization
     * Thrust dorsal
  2. - MCE:
     * Isometric contraction of the deep neck flexors.
     * Isometric contraction of the neck extensors.
     * Neural self-mobilization.
     * Cervical retraction with theraband.
     * Sphinx.
     * Scapular adduction exercises in prone.
     * Scapular adduction exercises in sitting position with theraband.
  Interventions: Other: IMT + Manual Therapy and Motor Control Exercise

INTERVENTIONS:
Other: Inspiratory Muscle training — This protocol will be performed using the Powerbreathe classic level 1 device and Yoga Respiratory Exercises (Pranayama)
  Arms: Inspiratory Muscle Training Group (IMT)
Other: IMT + Manual Therapy and Motor Control Exercise — The Inspiratory Muscle Training protocol will be performed using the Powerbreathe classic level 1 device and Yoga Respiratory Exercises (Pranayama). Manual Therapy and Motor Control Exercises will consist of joint mobilization/manipulation and exercises in the neck and thoracic regions
  Arms: IMT + Manual Therapy and Motor Control Exercises

SUMMARY:
The aim of this study is to assess if an intervention of manual therapy and motor control exercises combined with an inspiratory muscle training program is more effective than an inspiratory muscle training program alone in increasing the maximum inspiratory pressure in moderate smokers. In addition, the study pretends to evaluate the changes caused by the intervention regarding possible postural changes and thoracic diameter.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged between 18 and 60 years and a current smoking rate ≥ 5 points.

Exclusion Criteria:

* Were excluded participants who presented diagnosis of cardiorespiratory disease, systemic or metabolic disease such as rheumatoid arthritis or cancer, history of thoracic surgery, vertebral fracture, spinal structured musculoskeletal disorders and thoracic region and contraindication to the treatment techniques used (osteoporosis).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Maximum Inspiratory Pressure | Change from Baseline in Maximum Inspiratory Pressure at 4 weeks
  The maximum inspiratory pressure (MIP) was measured with a device called Kinetic KH1 Powerbreath (HAB International Ltd., England, UK). This device applies an inspiratory load which provides a resistance. The maneuver was performed in a sitting position. Measuring a minimum of 3 times was performed, recording the highest value.

SECONDARY OUTCOMES:
Head posture | Change from Baseline in Head Posture at 4 weeks
  The head posture was measured through the Cervical Range of Motion (CROM) device. This instrument measures physiological movements of the cervical spine and head position. It´s a reliable method of measuring, providing a range of intra-meter reliability from 0.7 to 0.9 and a range of inter-meter reliability from 0.8 to 0.87. The evaluator instructed the patient to sit in a standardized position and assume a natural position of the head and the goniometer was placed over his head to measure the head posture.
Thoracic kyphosis | Change from Baseline in Thoracic kyphosis at 4 weeks
  The measurement of the thoracic kyphosis was performed through flexicurve. It is a flexible rule that is molded to the back of the subject in order to replicate the shape of the spine. The flexicurve is a valid and reliable tool. The spinous processes of C7 and T12 were located, subsequently it placed on paper 10x10 to draw the curve and to obtained the index flexicurve.
Volumes and lung capacities | Change from Baseline in Volumes and lung capacities at 4 weeks
  The investigators used a simple Spirometry. The Spirometry was performed according to American Thoracic Society criteria with a portable Spirometer model spirobank usb (MIR Rome, Italy). The measures assessed in this outcome were: Forced Vital Capacity (FVC), Forced Expiratory Volume at the First second (FEV1), and Peak Expiratory Flow (PEF). The maneuver was performed 3 times and recording the best one

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Superior de Estudios Universitarios La Salle, Madrid, Madrid, Spain